CLINICAL TRIAL: NCT01297790
Title: Cough Responses to Tussive Agents in Health and Disease
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: JAS Protocol 2
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Obstructive Airway Disease; Asthma; Chronic Cough
Keywords: Cough; Inhalational cough challenges; Cough reflex sensitivity; Chronic cough.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Chronic Cough; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Asthma: Subjects with asthma more than 18 years old with minimal or no smoking history and evidence of bronchial hyperreactivity
  Interventions: Other: Cough Challenge Tests; Other: ambulatory cough recording; Other: Cough questionnaires
- Chronic obstructive pulmonary disease: Subjects with diagnosis of COPD who must be ex smokers and have evidence of airflow obstruction on breathing tests.
  Interventions: Other: Cough Challenge Tests; Other: ambulatory cough recording; Other: Cough questionnaires
- Healthy Volunteers: Healthy non smoking adults.
  Interventions: Other: Cough Challenge Tests; Other: ambulatory cough recording; Other: Cough questionnaires
- Healthy smokers: Current smokers with normal breath tests (spirometry)
  Interventions: Other: Cough Challenge Tests; Other: ambulatory cough recording; Other: Cough questionnaires
- Chronic cough: Subjects with idiopathic chronic cough.
  Interventions: Other: Cough Challenge Tests; Other: ambulatory cough recording; Other: Cough questionnaires

INTERVENTIONS:
Other: Cough Challenge Tests — Inhalational cough challenge tests with capsaicin, bradykinin, Citric acid and prostaglandin E2
Other: ambulatory cough recording — Cough recording with a portable device to capture cough sounds
Other: Cough questionnaires — Questionnaires designed to study cough. These include Leicester cough questionnaire, cough visual analogue score and cough quality of life questionnaire.

SUMMARY:
The sensitivity of a persons cough reflex can be measured by getting them to breath in (inhale) irritant chemicals. The purpose of this clinical research study is to test the sensitivity of the cough reflex to a variety of chemicals that can be inhaled to see if coughing responses are different between healthy people and people with respiratory problems that make them cough.

DETAILED DESCRIPTION:
Coughing is a distressing symptom which has a major impact on quality of life. It has been estimated that cough costs the UK economy £1 billion each year. Currently there are no effective anti-tussive agents to treat subjects with cough. Although drugs such as morphine may have some anti-tussive effect, side effects unacceptable.

Currently our understanding of the mechanisms which lead to coughing in different diseases is poor. Many mechanistic studies rely on testing the sensitivity of the cough reflex by inhalation of capsaicin (chilli-pepper extract) or citric acid. These challenges do not differentiate well between health and disease or between different disease states. Other agents such as prostaglandins and bradykinin are known to stimulate a coughing but responses to these agents have rarely been used as a measure of cough reflex sensitivity and not been compared to standard challenges.

It is clear that patients with common airway diseases such as COPD and asthma cough significantly more than healthy subjects. Moreover subjects presenting with chronic cough have cough rates an order of magnitude higher than most patients with airway disease. These differences are poorly represented by the differences in current cough challenge tests.

The investigators hypothesize that patterns of cough responses to different tussive agent may better differentiate between health and different disease states. These patterns may also suggest the different mechanisms leading to cough in different diseases.

ELIGIBILITY:
Inclusion Criteria:

* General

  * Adult subjects aged 18 years and over
  * Meet criteria for subject groups as outlined below

    (1) Healthy volunteers
  * Non-smokers
  * No history of respiratory disease

    (2) Healthy smokers
  * Current smokers with smoking history of ≥10 pack years
  * Spirometry within normal limits i.e. FEV1>80% predicted and FEV1/FVC ratio >75% predicted

    (3) Asthma
  * Physician diagnosis of asthma
  * Airways hyperresponsiveness to methacholine; PC20<16mg/ml (within last 2 years)
  * Non-smokers or ex-smoker with smoking history of ≤10 pack years

    (4) COPD
  * Physician diagnosis of COPD
  * Ex-smokers with smoking history of ≥20 pack years
  * Spirometry demonstrating airflow obstruction i.e. FEV1/FVC ratio <70%

    (5) Chronic Cough
  * History of a dry cough for >8 weeks
  * Normal CXR
  * Non-smokers or ex-smoker with smoking history of ≤10 pack years

Exclusion Criteria:

* 1) Symptoms of upper respiratory tract infection within the last 6 weeks 2) Participation in another clinical trial of an investigational drug within the last 4 weeks 3) Use of medication likely to alter cough reflex sensitivity i.e. ACE inhibitors, codeine phosphate, morphine sulphate, 4) Patients with severe respiratory disease i.e. FEV1 < 1 litre, 5) Significant medical co-morbidities likely to affect ability to participate in the trial or affect cough reflex sensitivity e.g. diabetes, stroke, Parkinson's disease, multiple sclerosis etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 and over who are healthy non smokers, or are current smokers with no respiratory conditions and normal spirometry, or have a diagnosis of asthma, chronic cough or COPD.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Cough response to tussive agents | 45 minutes
  To measure cough responses to capsaicin, citric acid, prostaglandin E2 (PGE2) and Bradykinin (BK) in healthy volunteers, airway diseases (asthma and COPD) and chronic cough.
  To compare the ability of individual challenges and patterns of challenge response to discriminate between diagnostic groups.
Objective cough recording | 24 Hours
  To perform ambulatory cough recording over 24 hours to assess if there are any differences

SECONDARY OUTCOMES:
C2 to inhaled tussive agents | 45 minutes
  C2 concentration difference between different diagnostic groups after inhalation of tussive agents

CONTACTS AND LOCATIONS:
Overall Officials: Ashley A Woodcock, FRCP, MD, Principal Investigator — University Hospital of South Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, Lancashire, United Kingdom

REFERENCES:
- [Derived] Belvisi MG, Birrell MA, Khalid S, Wortley MA, Dockry R, Coote J, Holt K, Dubuis E, Kelsall A, Maher SA, Bonvini S, Woodcock A, Smith JA. Neurophenotypes in Airway Diseases. Insights from Translational Cough Studies. Am J Respir Crit Care Med. 2016 Jun 15;193(12):1364-72. doi: 10.1164/rccm.201508-1602OC. PMID 26741046